CLINICAL TRIAL: NCT01812187
Title: Development of an Interactive, Adaptable and Transportable Treatment for Veterans With Substance Use Disorders
Brief Title: Designing a Mobile App for Veterans With Substance Use Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jan Lindsay, Ph.D., Principal Investigator, Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30374
Record Dates: First submitted 2013-03-04; First posted 2013-03-18 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Substance Abuse Problem; Alcohol Abuse; Alcohol Dependence
Keywords: Alcohol; Alcohol Abuse; Alcohol Dependence; Veterans
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHIFT Cognitive Behavioral Therapy (Experimental): Service to Home for Individually-Focused Therapy (SHIFT), a Cognitive Behavioral Treatment for Substance Use Disorders
  Interventions: Behavioral: SHIFT Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: SHIFT Cognitive Behavioral Therapy — Manualized, evidence-based, cognitive behavioral therapy for the treatment of substance abuse disorders
  Other Names: Service to Home for Individually Focused Therapy

SUMMARY:
The purpose of this study is to increase access for rural Veterans to evidence-based, person-centered, individually tailored treatment for alcohol use problems. The primary aim is to evaluate the acceptability and feasibility of using mobile technology deliver treatment for alcohol use disorder. A mobile application will be used replacing the usual setting of clinical visits that accompanies standard face-to-face CBT therapy. The application will be loaded onto an iPod, which will be distributed to each participant that has been found to be eligible to participate.

DETAILED DESCRIPTION:
Many Veterans returning from Iraq and Afghanistan experience problems with drinking. There are treatments for alcohol use disorders that can be very helpful, but sometimes it can be hard for Veterans to find or participate in the treatments. This can be because of the amount of time the treatments take and the long distance to places where substance abuse treatments are offered. For Veterans who live in rural areas, these types of issues can pose even bigger problems. To address these issues, new types of treatments and ways of delivering care are being studied.

We have developed a mobile application that will be accessed through the use of a mobile device such as an ipod. The application will contain an application dedicated to the treatment of substance abuse disorders. This application will provide the coping skills and educational information to aide in helping with problems associated with drinking alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran of the Armed Forces
2. are part of the primary care - mental health (PC-MH)
3. reside in a rural community, as defined by the US Census Bureau
4. score greater than or equal to 8 on the Alcohol Use Disorder Identification Test (AUDIT)
5. meet diagnostic criteria for alcohol abuse or dependence as assessed by the Mini International Neuropsychiatric Inventory (MINI) according to the Diagnostic and Statistical Manual (DSM-IV)
6. Age 18 and older to participate. -

Exclusion Criteria:

1. Have conditions that threaten your safety (e.g., active suicidal intent, current uncontrolled psychosis or bipolar disorders in the past month as assessed by the MINI).
2. Veterans with a diagnosed concurrent substance dependence (other than nicotine) and more than mild risk of alcohol withdrawal based on a score of greater than 8 on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA-Ar) will be excluded.

   -

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change | Change from baseline AUDIT score at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Lindsay, Ph.D., Principal Investigator — Baylor College of Medicine; Michael E. Debakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States